CLINICAL TRIAL: NCT05278403
Title: Use of Virtual Reality and Video Games in the Physiotherapy Treatment of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Angel Martínez Carrasco, Professor Phd, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JPV-2022-01
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Stroke; Virtual Reality; Physical Therapy
MeSH Terms: conditions — Stroke | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Two randomized groups. A control group and an experimental group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomized groups. Participants do not know to which group they are assigned. The other participants are unaware of the purpose of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Conventional neurological physiotherapy treatment.
  Interventions: Other: Neurological physiotherapy
- Experimental group (Experimental): Conventional neurological physiotherapy treatment with the use of virtual reality and video games.
  Interventions: Other: Virtual reality and video games; Other: Neurological physiotherapy

INTERVENTIONS:
Other: Virtual reality and video games — Use of a software in stroke patients' rehabilitation.
  Arms: Experimental group
Other: Neurological physiotherapy — Application of conventional physical therapy techniques.

SUMMARY:
Randomized clinical trial based on the application of virtual reality and video games together with physiotherapy treatment in stroke patients, with the main objective of determining their beneficial effects.

DETAILED DESCRIPTION:
21 participants who will be divided by randomization between a control group and an experimental group. The results will be quantified with the following scales: Modified Asworth (spasticity). Daniels et al (muscle strength) Tinetti (balance and gait) Berg (balance) Joint range

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving neurological physiotherapy treatment.
* Patients who have suffered a stroke in the last two years.
* Patients with an age range between 18 and 80 years old.
* Patients with stroke with the ability to have minimal manual pressure with one limb.

Exclusion Criteria:

* Patients with stroke who also have degenerative diseases such as Alzheimer's or Parkinson's.
* Stroke patients who do not understand the instructions.
* Patients who have undergone surgery on the evaluated limbs.
* Patients with scars that limit movement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
Strength | One month
  Strength measurement using the Daniels and Worthingham Scale. Minimum value = 0 , maximum value = 5. Higher scores mean a better outcome.
Spasticity | One month
  Spasticity measurement using the Ashworth modified scale. Minimum value = 0, maximum value = 4. Higher scores mean a worse outcome.
Gait | One month
  Gait measurement using the Tinetti scale. Minimum value = 0, maximum value = 28. Higher scores mean a better outcome.
Balance | One month
  Balance using the Berg Balance Scale. Minimum value = 0, maximum value = 56. Higher scores mean a better outcome.
Joint range | One month
  Joint range measure using goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Angel Martínez Carrasco, PhD, Study Director — Universidad de Murcia; Francisco Javier Peláez Vélez, Graduated, Principal Investigator — Universidad de Murcia
Locations (1):
- Universidad de Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No